CLINICAL TRIAL: NCT03910998
Title: A Randomized Parallel Design Study to Compare the Impact of Intraoperative Deep Neuromuscular Blockade on Intraoperative NOL-guided Opioid Requirement and Postoperative Early Outcomes in Laparoscopic Colorectal Surgeries
Brief Title: Impact of Intraoperative Deep Neuromuscular Blockade on NOL-guided Opioid Requirement in LSC Colorectal Surgeries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ciusss de L'Est de l'Île de Montréal (Other)
Collaborators: Merck Canada Inc. (Industry)
Responsible Party: Principal Investigator, Philippe Richebe, Director of Research, Principal Investigator, Anesthesiologist, Associate Professor, MD, PhD, Ciusss de L'Est de l'Île de Montréal
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-1610
Record Dates: First submitted 2019-03-04; First posted 2019-04-10 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Laparoscopic Colorectal Surgeries
Keywords: neuromuscular blockade; NOL monitoring; opioid consumption; intraoperative; anesthesia

STUDY DESIGN:
Intervention Model Description: Tow groups of patients. Randomization into group "D" for Deep muscle relaxation vs group "M" for Moderate muscle relaxation according to a randomization list for a total number of 100 patients
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization into group "D" for Deep muscle relaxation (high doses of intraoperative rocuronium and antagonization at the end with 4mg/kg of suggamadex) vs group "M" for Moderate muscle relaxation (moderate doses of intraoperative rocuronium and antagonization at the end with suggamadex 2mg/kg) will be done prior to the entrance in the OR, the day of the surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group "M" for Moderate muscle relaxation, low doses rocuronium (Active Comparator): A bolus of 0.4 mg/kg of IV rocuronium will be given at the induction of the anesthesia.
  Rocuronium IV bolus guided by TOF that must remain between 1-3 / 4 during surgery.
  Interventions: Drug: Rocuronium IV bolus 0.1 mg/kg guided by TOF that must remain between 1-3 during surgery
- Group "D" for Deep muscle relaxation, high doses rocuronium (Experimental): A bolus of 0.4 mg/kg of IV rocuronium will be given at the induction of the anesthesia.
  Bolus of rocuronium 0.1 mg/kg IV will be given during surgery to keep the TOF 0/4 and a PTC ≤ 2 (parameters measured every 10 minutes).
  Interventions: Drug: Rocuronium IV bolus 0.1 mg/kg guided by TOF 0/4 and PTC≤ 2

INTERVENTIONS:
Drug: Rocuronium IV bolus 0.1 mg/kg guided by TOF that must remain between 1-3 during surgery — Bolus of rocuronium 0.1 mg/kg at the discretion of anesthetist to keep the TOF between 1-3 out of 4 during surgery
  Arms: Group "M" for Moderate muscle relaxation, low doses rocuronium
Drug: Rocuronium IV bolus 0.1 mg/kg guided by TOF 0/4 and PTC≤ 2 — Bolus of rocuronium 0.1 mg/kg IV will be given during surgery for a TOF 0/4 and a PTC ≤ 2 (parameters measured every 10 minutes).
  Arms: Group "D" for Deep muscle relaxation, high doses rocuronium

SUMMARY:
The aim of the present study is to answer the question whether deep neuromuscular blockade has a clinically significant impact on intra and postoperative pain, opioid requirement and anesthesia related outcomes and side effects for the early phase of recovery (24hs) after colorectal laparoscopic surgery.

DETAILED DESCRIPTION:
Background: For the last decade many studies have reported that intraoperative surgical and anesthesia conditions might have an impact of postoperative pain.

The most recent surgical literature agrees on the fact the IAP should remain under 15mmhg or even 12mmhg during the whole laparoscopic surgery, and many efforts to do so were developed in the most recent years. On the anesthesia side, deep neuromuscular block was associated with better postoperative recovery when looking at pain parameters such as pain scores and opioid requirements. Nevertheless, all these previous studies, even if recent, did not properly evaluate intraoperative pain and did not well control criteria used to guide the administration of intraoperative opioids, one of the main components of anesthesia. Also, lots of these studies did not properly evaluate or control the depth of hypnosis, another main component of anesthesia. Nowadays, new monitors with extremely better sensitivity and specificity are available for each of the anesthesia component. This might completely revisit the previous findings in the literature and offer much better-quality results. Maisonneuve-Rosemont Hospital in Montreal is a unique center that has invested in new monitors to evaluate each of these anesthesia component: BIS index for depth of hypnosis (BIS device, Covidien, Saint-Laurent, Canada), NOL index (PM-200TM device, Medasense LTD, Ramat Gan, Israel) for nociceptive evaluation (intra-operative pain assessment under general anesthesia), and TOF-scan (NMB monitor, Drager, Mississauga, Canada) for quantitative and 3D evaluation of the depth of muscle relaxation.

This study will answer the question whether deep neuromuscular blockade has a clinically significant impact on intra and postoperative pain, opioid requirement and anesthesia related outcomes and side effects for the early phase of recovery (24hs) after colorectal laparoscopic surgery.

This study will be conducted in a single center, and will be an open label, single blinded, randomized controlled study. Type of surgery: laparoscopic colorectal surgery with anesthesia time expected to last more than 120min in ASA 1-3 patients, fully consented for primary colorectal laparoscopic surgery.

The primary objective of the study: To compare total intra-operative remifentanil consumption during anesthesia for laparoscopic colorectal surgery between two groups: Group "D" for Deep muscle relaxation and group "M" for Moderate muscle relaxation. Secondary objectives are listed below. For an expected decrease of 25% in the remifentanil intraoperative consumption per hour of surgery (in mcg) of surgery, with a type I error α = 0.05 (two-tailed), a 90% power, the total sample size needed is 82 (41 per group). To account for an approximative 20% rate of loss to follow-up or missing data due to technical problems, a total of 100 subjects will be recruited.

Study Duration: 24 months. Study Center: Maisonneuve-Rosemont Hospital, CIUSSS de l'Est de l'Ile de Montreal (CEMTL), University of Montreal, Montreal, Quebec, Canada.

Adverse Events: None expected. Subvention: An Independent Investigator Initiated Trial (IIIT) grant application has been accepted by the company Merck (see letter attached) for the sponsoring of this study.

ELIGIBILITY:
Inclusion Criteria:

* ASA1-3 patients,
* fully consented,
* primary colorectal laparoscopic surgery and no previous laparotomy for the last 5 years
* BMI < 35,
* Age > 18yo,
* no allergy to any of the medications used in this study.

Exclusion Criteria:

* history of coronary artery disease
* serious cardiac arrhythmia (including atrial fibrillation)
* history of substance abuse
* chronic use of psychotropic and/or opioid drugs
* use of drugs that act on the autonomic nervous system (including β-blockers)
* history of psychiatric diseases with the need of medication
* allergy to any drug used in the study protocol
* refusal of the patient for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Total intra-operative remifentanil consumption during surgery in mcg/kg/h | Intra-operative (from T0 incision until Tend = start dressing)
  To compare total intra-operative remifentanil consumption (in mcg per hour from T0 incision until Tend = start dressing) during anesthesia for laparoscopic colorectal surgery between two groups: Group "D" for Deep muscle relaxation and group "M" for Moderate muscle relaxation

SECONDARY OUTCOMES:
Number of IV boluses and increases of remifentanil infusion, number, no unit | Intra-operative (from T0 incision until Tend = start dressing)
  To compare the number of IV boluses and increases of remifentanil infusion needed in group D versus M
Number of times NOL index passes over the threshold of 25, number, no unit | Intra-operative (from T0 incision until Tend = start dressing)
  To compare the number of times NOL index passes over the threshold of 25 (considered as painful threshold in an anesthetized patient) during anesthesia in group D versus M
Area Under the Curve (AUCs) whenever the NOL is above 25, no unit | Intra-operative (from T0 incision until Tend = start dressing)
  To compare the Area Under the Curve (AUCs) of all the intraoperative periods for which the NOL index will be above the pain threshold of 25 from T0 until Tend
Total intraoperative time from T0 until Tend with NOL above 25 in minutes | Intra-operative (from T0 incision until Tend = start dressing)
  To compare the total intraoperative time in minutes from T0 until Tend with NOL index above 25, with NOL index between 10 and 25, and with NOL index below 10 in group D versus M
Intraoperative level of intra-abdominal pressure (IAP) in mmHg | Intra-operative (from T0 incision until Tend = start dressing)
  To compare between group D versus M the intraoperative level of intra-abdominal pressure (IAP) to keep a surgeons' satisfaction score (Leiden Surgical Rating Scale L-SRS)
Abdominal insufflation duration in minutes | Intra-operative (from T0 incision until Tend = start dressing)
  To compare the time in minutes spent with abdominal insufflation and laparoscopic surgery between group D and M
Time for awakening and extubation in seconds | Intra-operative (from T0 incision until Tend = start dressing)
  To compare the time for awakening and extubation (performed for all patients in the Operating Room, OR) between group D and M
Pain score at rest on a scale from 0 to 10 | every 15 minutes until discharge from PACU, up to 3 hours
  To compare maximal postoperative pain scores (Numeric Rating Scale, NRS) at: arrival in postanesthesia care unit (PACU), and every 15 min until PACU discharge at rest and coughing/mobilization
Pain score at coughing/mobilization on a scale from 0 to 10 | every 15 minutes until discharge from PACU, up to 3 hours
  To compare maximal postoperative pain scores (Numeric Rating Scale, NRS) at: arrival in postanesthesia care unit (PACU), and every 15 min until PACU discharge at rest and coughing/mobilization
Pain score at the shoulder on a scale from 0 to 10 | every 15 minutes until discharge from PACU, up to 3 hours
  To compare the incidence of shoulder pain and intensity (maximal NRS score at the shoulder) in PACU at arrival then every 15 minutes, between group D versus M
Postoperative Hydromorphone consumption in mg in Postoperative Care Unit (PACU) | every 15 minutes until discharge from PACU, up to 3 hours
  To compare the total amount of hydromorphone (in mg) given IV in PACU as a pain killer titration following a strict PACU protocol to reach a NRS pain score < 4/10 between group D and M
Pain score at rest at 8hs on a scale from 0 to 10 | 8 hours after surgery in hospital
  To compare maximal postoperative pain scores at rest at 8 hours after surgery between group D and M
Pain score at coughing/mobilization at 8hs on a scale from 0 to 10 | 8 hours after surgery in hospital
  To compare maximal postoperative pain scores at coughing/movement at 8 hours after surgery between group D and M
Pain score at rest at 16hs on a scale from 0 to 10 | 16 hours after surgery in hospital
  To compare maximal postoperative pain scores at rest at 16 hours after surgery between group D and M
Pain score at coughing/mobilization at 16hs on a scale from 0 to 10 | 16 hours after surgery in hospital
  To compare maximal postoperative pain scores at coughing/movement at 16 hours after surgery between group D and M
Pain score at rest at 24hs on a scale from 0 to 10 | 24 hours after surgery in hospital
  To compare maximal postoperative pain scores at rest at 24 hours after surgery between group D and M
Pain score at coughing/mobilization at 24hs on a scale from 0 to 10 | 24 hours after surgery in hospital
  To compare maximal postoperative pain scores at coughing/movement every 24 hours after surgery between group D and M
Amount of opioids received in 24h as Patient Controlled Analgesia in mg | 24 hours after surgery in hospital
  To compare analgesic requirements for 24 hours given as patient controlled analgesia (PCA) in mg over 24hs
Recovery score QOR15 questionnaire (150 points maximum for this questionnaire) | 24 hours after surgery in hospital
  To compare recovery scores (QOR15) from 0 to 150 points at 24 hours after surgery
POSS postoperative Sedation score in PACU on a scale from 1 to 4 | every 30 minutes from T0 = arrival in PACU until discharge from PACU, up to 3 hours
  Sedation score in PACU
postoperative nausea and vomiting score in PACU on a scale from 0 to 3 | every 30 minutes from T0 = arrival in PACU until discharge from PACU, up to 3 hours
  nausea and vomiting score in PACU from 0 to 3
postoperative Aldrete score in PACU on a scale from 5 to 15 | every 30 minutes from T0 = arrival in PACU until discharge from PACU, up to 3 hours
  Recovery score in PACU to decide on the possibility of discharge of the patient from PACU

CONTACTS AND LOCATIONS:
Overall Officials: Philippe PR Richebé, MD PhD, Principal Investigator — CIUSSS Est de l'île de Montréal
Locations (1):
- Hopital Maisonneuve Rosemont, CIUSSS de l'Est de l'Ile de Montréal, Montreal East, Quebec, Canada

REFERENCES:
- [Derived] Morisson L, Harkouk H, Othenin-Girard A, Oulehri W, Laferriere-Langlois P, Belanger ME, Idrissi M, Godin N, Verdonck O, Fortier LP, Poirier M, Henri M, Latulippe JF, Tremblay JF, Trepanier JS, Bendavid Y, Raft J, Richebe P. Impact of deep neuromuscular blockade on intraoperative NOL-guided remifentanil requirement during desflurane anesthesia in laparoscopic colorectal surgeries: A randomised controlled trial. J Clin Anesth. 2024 Dec;99:111659. doi: 10.1016/j.jclinane.2024.111659. Epub 2024 Oct 23. PMID 39447530